CLINICAL TRIAL: NCT02573025
Title: An Open-Label, Randomized, Multi-Center, Single Dose, Two-Period, Two Sequence Crossover Study to Investigate the Bioequivalence of Peginterferon (PEG-IFN) Alfa-2a Benzyl Alcohol-Free Formulation Versus the Reference Market Formulation Following Subcutaneous Administration Via Prefilled Syringe in Healthy Chinese Subjects
Brief Title: A Bioequivalence Study of Pegylated Interferon Alfa-2a (PEG-IFN Alfa-2a) Benzyl Alcohol (BA)-Free Formulation Versus PEG-IFN Alfa-2a (Pegasys) Following Subcutaneous Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: YV29573
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — peginterferon alfa-2a

ARMS (2):
- Test Followed by Reference (Experimental): Participants will receive PEG-IFN alfa-2a BA-free formulation (Test) in Period 1, followed by PEG-IFN alfa-2a market formulation (Reference) in Period 2 on Day 1 of each period with a washout period of 14 to 21 days.
  Interventions: Drug: PEG-IFN alfa-2a BA-free formulation (Test); Drug: PEG-IFN alfa-2a market formulation (Reference)
- Reference Followed by Test (Experimental): Participants will receive PEG-IFN alfa-2a market formulation (Reference) in Period 1, followed by PEG-IFN alfa-2a BA-free formulation (Test) in Period 2 on Day 1 of each period with a washout period of 14 to 21 days.
  Interventions: Drug: PEG-IFN alfa-2a BA-free formulation (Test); Drug: PEG-IFN alfa-2a market formulation (Reference)

INTERVENTIONS:
Drug: PEG-IFN alfa-2a BA-free formulation (Test) — Participants will receive single injection of 180 micrograms (mcg) of PEG-IFN alfa-2a BA-free formulation, subcutaneously via prefilled syringe in either period 1 and 2 (each period having 35 days).
Drug: PEG-IFN alfa-2a market formulation (Reference) — Participants will receive single injection of 180 mcg of PEG-IFN alfa-2a market formulation, subcutaneously via prefilled syringe in either period 1 and 2 (each period having 35 days).
  Other Names: Pegasys

SUMMARY:
This is an open-label, randomized, multi-center, single dose, two-period, two-sequence crossover study to investigate the bioequivalence of PEG-IFN alfa-2a BA-free formulation versus the reference market formulation (PEG-IFN alfa-2a [Pegasys®]) following subcutaneous administration via prefilled syringe in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male Chinese participants
* Body mass index between 19 and 28 kilograms per square meter (kg/m^2), inclusive
* Participants determined as healthy by their medical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory measurements performed at the Screening visit
* Female participants of childbearing potential: willing to use highly effective methods of contraception throughout the study and for 90 days after the last dosing
* Male participants: agreement to remain abstinent or use spermicide and barrier method contraception throughout the study and for 90 days after the last dosing
* Able to participate and willing to give written informed consent and to comply with the study restrictions

Exclusion Criteria:

* Any clinically relevant condition or history of cardiovascular, psychiatric, gastrointestinal, respiratory, renal, hepatic, hematological, lymphatic, neurological (including seizure history), musculoskeletal, genitourinary, immunological, metabolic, malignant, or dermatological disorder
* Participants who are positive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti HCV) or human immunodeficiency virus I and II antibody (anti-HIV I, anti-HIV II) tests at Screening
* Participants with alanine aminotransferase (ALT) above the upper limit of normal at Screening or on Day -1 of Period 1
* Any other condition or disease (other than those already stated) which, in the judgment of the Investigator, would place the participant at undue risk, interfere with the absorption, distribution, metabolism, and excretion of PEG-IFN alfa-2a, or interfere with the ability of the participant to complete the study
* History of drug or alcohol abuse within the last year before screening
* Treatment with interferon or PEG-IFN alfa-2a within 3 months prior to the first dosing
* Female participants who are pregnant, currently lactating, or have a positive serum pregnancy test at screening or have a positive urine pregnancy test on Day -1 of Period 1
* Use of any prescribed or over the counter medication or herbal medicine taken within 14 days prior to the first dosing or within 5 times the elimination half-life of the medication prior to the first dosing (whichever is longer). Exceptions are paracetamol, the contraceptive pill, hormone replacement therapy and commonly used vitamin supplements, which are permitted
* Regular smoking with consumption of more than 10 cigarettes per day or an equivalent amount of tobacco
* Participation in an investigational drug or device study within 3 months prior to the first dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2016-04-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) for PEG-IFN alfa-2a | Predose (-1 Hour), Hour 1, 3, 5, 8, 12, 24, 48, 72, 84, 96, 120, 144, 168, 192, 216, 240, 312, 384, 480, 552, 648, 816 post Dose
Area Under the Concentration-Time Curve (AUC) for PEG-IFN alfa-2a From Time Zero to 816 hours (AUC0-816h) | Predose (-1 Hour), Hour 1, 3, 5, 8, 12, 24, 48, 72, 84, 96, 120, 144, 168, 192, 216, 240, 312, 384, 480, 552, 648, 816 post Dose

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve for PEG-IFN alfa-2a From Time Zero Extrapolated to Infinity (AUC0-inf) | Predose (-1 Hour), Hour 1, 3, 5, 8, 12, 24, 48, 72, 84, 96, 120, 144, 168, 192, 216, 240, 312, 384, 480, 552, 648, 816 post Dose
Time to Reach Cmax (tmax) for PEG-IFN alfa-2a | Predose (-1 Hour), Hour 1, 3, 5, 8, 12, 24, 48, 72, 84, 96, 120, 144, 168, 192, 216, 240, 312, 384, 480, 552, 648, 816 post Dose
Terminal Half-Life (t1/2) for PEG-IFN alfa-2a | Predose (-1 Hour), Hour 1, 3, 5, 8, 12, 24, 48, 72, 84, 96, 120, 144, 168, 192, 216, 240, 312, 384, 480, 552, 648, 816 post Dose
Percentage of Participants With Adverse Events | Baseline up to 35 days post last dose of PEG-IFN alfa-2a (maximum up to 17.5 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- CMAX A division of IDT Australia Limited, Adelaide, South Australia, Australia
- Hong Kong (2):
  - The University of Hong Kong; Pharmacy Clinical Trials, Hong Kong
  - The Chinese University of Hong Kong; Emergency Medicine, Shatin
- New Zealand (2):
  - Christchurch Clinical Studies Trust, Christchurch
  - Auckland Clinical Studies Limited, Grafton
- Singapore (2):
  - SingHealth Investigational Medicine Unit; Haematology, Singapore
  - Changi General Hospital- Parent; Department of Rheumatology, Singapore
- Taiwan (2):
  - China Medical University Hospital;Oncology and Hematology Office Critical Care Center, 14H, Taichung
  - Taipei Medical University Hospital; Clinical Research Center, Taipei